CLINICAL TRIAL: NCT04994444
Title: Preloading With Nicotine Replacement Therapy in HIV-positive Smokers to Improve Self-Efficacy and Quit Attempts
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2102002917; 1R21CA261233-01 (NIH)
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use Cessation
Keywords: smoking; HIV; Cessation
MeSH Terms: conditions — Tobacco Use Cessation; Smoking | interventions — Nicotine; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The Research Assistant collecting data at assessment sessions will not be aware of the participant's study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Preloading (Experimental): Participants will be started on nicotine patch 3 weeks prior to quit date. At quit date they will use patch and lozenge or gum for 8 weeks.
  Interventions: Drug: Nicoderm CQ 21Mg/24Hr Transdermal System
- Standard treatment (Active Comparator): Participants will start combination nicotine replacement therapy (patch/gum or patch/lozenge) on their assigned quit date. NRT will be provided for 8 weeks.
  Interventions: Drug: Nicoderm CQ 21Mg/24Hr Transdermal System

INTERVENTIONS:
Drug: Nicoderm CQ 21Mg/24Hr Transdermal System — Nicoderm CQ patch started 3 weeks prior to quit date. Starting on quit date, patch/gum or patch/lozenge will be used for 8 weeks. Patch will be tapered over the 8 week period.
  Other Names: Nicotine replacement therapy

SUMMARY:
The overall goal of this research project is to examine the feasibility, acceptability, and preliminary efficacy of nicotine replacement therapy preloading (NRT-P) in HIV-positive smokers, who are struggling with cigarette dependence, urge to smoke (craving) and low self-efficacy as barriers to successful smoking cessation. Sixty participants will be recruited into a 16-week randomized pilot study. Thirty participants (control condition) will receive standard smoking cessation counseling (NRT-S) and will initiate an 8-week course of combination nicotine patch and lozenge (or gum, based on preference) on quit date (week 4), consistent with recommended guidelines based on smoking rate. Thirty participants (active condition) will start NRT patch 3 weeks prior to quit date, followed by an 8-week course of combination nicotine patch and lozenge (or gum, based on preference), initiated on quit date. The investigators will examine dependence, urge to smoke and self-efficacy for quitting prior to and following quit date. The investigators will also examine differences in quit attempts and biochemically validated smoking abstinence between the control and active conditions at weeks 8, 12, and 16.

DETAILED DESCRIPTION:
Cigarette smoking is more prevalent in persons with HIV (PWH) in the U.S. when compared with the general population and is linked to increased morbidity and mortality in this population. Furthermore, HIV-positive smokers have increased rates of lung and other smoking-related cancers. Smokers with HIV are a particularly challenging group, often reporting high severity of nicotine dependence and low rates of self-efficacy for quitting, both factors related to poor smoking cessation outcomes. Establishing more effective smoking cessation approaches for smokers with HIV, particularly those that address low self-efficacy and severe dependence, is a public health priority. The overall goal of this research project is to examine the feasibility, acceptability, and preliminary efficacy of nicotine replacement therapy preloading (NRT-P) in HIV-positive smokers, who are struggling with cigarette dependence, urge to smoke (craving) and low self-efficacy as barriers to successful smoking cessation. Sixty participants will be recruited into a 12-week randomized pilot study. Thirty participants (control condition) will receive standard smoking cessation counseling (NRT-S) and will initiate an 8-week course of combination nicotine patch and lozenge on quit date (week 4), consistent with recommended guideline based on smoking rate. Thirty participants (active condition) will start NRT patch 3 weeks prior to quit date, followed by an 8-week course of combination nicotine patch and lozenge, initiated on quit date. Dependence, urge to smoke and self-efficacy for quitting prior to and following quit date will be examined. Differences in quit attempts and biochemically validated smoking abstinence between the control and active conditions at weeks 8 and 12 will also be examined. This study will be the first to examine the feasibility and initial efficacy of a novel intervention using NRT preloading to improve smoking cessation outcomes in PWH. Given the high prevalence of smoking and the significant morbidity associated with it in PWH, the development of effective strategies to reduce the risks related to smoking in this group is critical. If determined to be effective, this intervention could be readily disseminated in HIV clinics. This study will provide key information on the potential benefit of NRT preloading in a population that is highly dependent on nicotine and highly vulnerable to smoking-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with HIV
* at least 18 years of age
* smoking at least 5 cigarettes/day
* exhaled Carbon Monoxide level greater than 5 at baseline
* willing to use transdermal nicotine patch
* ready to quit in the next 30 days.

Exclusion Criteria:

* currently using pharmacotherapy for smoking cessation
* medically or psychiatrically unstable (defined as: uncontrolled hypertension, unstable angina, or a medical or psychiatric hospitalization in the 30 days prior to enrollment) *experiencing psychotic symptoms
* endorsing suicidal ideation upon screening or past-year suicide attempt
* pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Cioe, PhD, Principal Investigator — Brown University School of Public Health
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will include data from 60 subjects being enrolled into a pilot randomized clinical trial where participants who smoke combustible cigarettes will be randomized to one of two conditions: the nicotine replacement therapy preloading condition (NRT-P), or the standard treatment condition (ST). The final dataset will include self-reported demographic and behavioral data from interviews with the subjects. The final dataset will be stripped of identifiers prior to release for sharing. We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preloading | Standard Treatment
Started | 23 | 26
Completed | 19 | 20
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preloading | Standard Treatment | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (14.1) | 52.0 (11.5) | 52.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 9 | 8 | 17
  sex: Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 7 | 12
  White | 16 | 15 | 31
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 26 | 49
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] | 14.1 (8.6) | 15.5 (9.8) | 14.9 (9.2)
Years of smoking cigarettes [Mean (Standard Deviation); unit: years] | 32.2 (16.5) | 30.0 (14.7) | 31.0 (15.5)
Fagerstrom test of cigarette dependence (FTCD) [Mean (Standard Deviation); unit: units on a scale] — the FTCD measures cigarette dependence. The scale has 6 items and scores are added for a total score. The overall score can range from 0 (no dependence) to 10 (high dependence). Higher scores indicate higher dependence on cigarettes.
  units on a scale | 4.7 (2.0) | 4.9 (2.6) | 4.8 (2.3)
Confidence to Quit [Mean (Standard Deviation); unit: units on a scale] — The Confidence to quit scale is a 1-item scale that asks, "On a scale of 1 to 10, how confident are you that you would be able to quit smoking cigarettes permanently'? Range 1 to 10, with 1="not at all confident" and 10= "completely confident"
  units on a scale | 7.2 (2.3) | 7.2 (2.0) | 7.2 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Adherence to NRT
Description: Number of days of nicotine patch use during the 8 weeks of provision
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: days of NRT use
Arm/Group | Preloading | Standard Treatment
Number analyzed (Participants) | 23 | 26
days of NRT use | 47.4 (13.2) | 32.7 (21.8)

2. Secondary Outcome: 7 Day Point Prevalence Abstinence
Description: number of participants who reported no cigarette smoking in past 7 days
Time Frame: week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Preloading | Standard Treatment
Number analyzed (Participants) | 23 | 26
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Preloading | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT04994444/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT04994444/ICF_001.pdf